# ClinicalTrials.gov Study Protocol

Official Title: Diastolic Dysfunction in the Pregnant Woman with Preeclampsia: A Prospective Observational Study at the Maternity and Neonatology Center of Tunis

Short Title: Diastolic Dysfunction in Preeclampsia

NCT Number: [to be assigned]

Date: August 2025

Sponsor/Responsible Party: Maternity and Neonatology Center of Tunis

Principal Investigator: [DR Sarra zarrouk, MD, Maternity and Neonatology Center of Tunis,

Tunisia, zarrouk.sarah958@gmail.com]

## 1. Objective

The objective of this study is to evaluate diastolic function in pregnant women with preeclampsia and to compare findings with normotensive pregnant women.

## 2. Study Design

- Study Type: Observational (Case-Control)
- Study Model: Case-Control, two cohorts (Preeclampsia vs. Normotensive)
- Time Perspective: Prospective
- Enrollment: 80 participants (40 in each cohort)
- Follow-up Duration: Until delivery and immediate postpartum (up to 7 days)

## 3. Study Setting and Duration

This study was conducted within the Anesthesia-Resuscitation and Gynecology-Obstetrics Departments (A, B, C, and D) of the Maternity and Neonatology Center in Tunis, Tunisia, over a 5-month period from March 2025 to June 2025.

## 4. Eligibility Criteria

Inclusion Criteria:

- Pregnant women aged 18-45 years
- Third trimester of pregnancy
- Group A: women diagnosed with preeclampsia (≥140/90 mmHg after 20 weeks + proteinuria ≥300 mg/24h, with or without severity criteria)
- Group B: normotensive pregnant women without proteinuria (<300 mg/24h if tested)

#### **Exclusion Criteria:**

- Pre-existing cardiovascular disease (valvulopathy, cardiomyopathy, EF <50%)
- Congenital heart disease, arrhythmia, prior cardiac surgery
- Chronic hypertension (before 20 weeks)
- Pulmonary hypertension (pre- or post-capillary)
- Systemic disease with cardiac involvement (SLE, Behçet's disease)
- Technical difficulty preventing echocardiographic evaluation
- Unusable medical records or diagnostic uncertainty
- Gestational hypertension without preeclampsia

# 5. Study Procedures

## Data Collection:

- Demographics, medical history, clinical and biological data collected using standardized forms.
- Echocardiographic parameters recorded according to ASE/EACVI 2016 guidelines.

Echocardiographic Parameters Assessed:

- Transmitral Doppler flow (E wave, A wave, E/A ratio, Deceleration Time)
- Tissue Doppler imaging (E' septal, E' lateral, A', S')
- Indexed left atrial volume
- Maximum tricuspid regurgitation velocity (Vmax TR)

#### Classification of Diastolic Function:

- Normal
- Indeterminate
- Diastolic Dysfunction (Grade I = impaired relaxation; Grade II = pseudonormal; Grade III = restrictive)

#### 6. Outcome Measures

#### **Primary Outcome:**

- Title: Prevalence of left ventricular diastolic dysfunction in preeclamptic women
- Description: Echocardiographic evaluation based on ASE/EACVI 2016 criteria
- Time Frame: At echocardiographic evaluation during the third trimester

## **Secondary Outcomes:**

- 1. Comparison of diastolic parameters between preeclamptic and normotensive groups (E', E/E', LA volume, TR velocity).
- 2. Association between diastolic dysfunction and maternal symptoms (dyspnea, palpitations, pulmonary edema).
- 3. Correlation between severity of preeclampsia and degree of diastolic dysfunction.
- Time Frame: During pregnancy and up to 7 days postpartum.

## 7. Statistical Analysis Plan

- Continuous variables expressed as mean  $\pm$  SD; compared using Student's t-test or Mann-Whitney U test.
- Categorical variables expressed as counts (%) and compared using Chi-square or Fisher's exact test.
- p < 0.05 considered statistically significant.
- Subgroup analysis: association between severity of preeclampsia and prevalence of diastolic dysfunction.

#### 8. Ethical Considerations

- Study approved by the Local Ethics Committee of the Maternity and Neonatology Center of Tunis.

- Written informed consent obtained from all participants.
- Confidentiality, anonymity, and protection of personal data ensured.

# 9. References

ASE/EACVI 2016 Guidelines on Diastolic Function. Melchiorre K et al. Circulation. 2011. Guirguis G et al. J Am Soc Echocardiogr. 2015.